CLINICAL TRIAL: NCT07306806
Title: Comparison of Post-Operative Analgesia of Caudal Versus Dorsal Penile Nerve Blocks for Pediatric Patients Undergoing Hypospadias Repair
Brief Title: Caudal vs Dorsal Penile Nerve Block for Postoperative Analgesia in Children Undergoing Hypospadias Repair (CaD-DPNB)
Acronym: CaD-DPNB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Kamal Habib, Lecturer of Anesthesiology and Critical Care, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMASU MS 575/ 2021
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Hypospadias Repair; Pediatric Anesthesia; Postoperative Analgesia
Keywords: DPB vs caudal block in hypospadius repair

STUDY DESIGN:
Intervention Model Description: This study follows a randomized parallel-group interventional model comparing two established regional anesthesia techniques: caudal block and dorsal penile nerve block. Participants are randomly allocated in a 1:1 ratio using concealed assignment to ensure unbiased group distribution. Each participant receives only the technique assigned, with no crossover permitted. Standardized protocols are applied for induction, drug dosing, positioning, and monitoring to minimize procedural variability. Outcome assessors and data collectors are blinded to group allocation whenever feasible. Both groups follow identical perioperative timelines, including preoperative evaluation, intraoperative monitoring, and postoperative pain assessment. This model allows a controlled and unbiased comparison of the efficacy, safety, and clinical performance of the two techniques under uniform conditions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal epidural block (Experimental): Participants receive a single caudal epidural injection of 0.25% bupivacaine (0.5 mL/kg) via the sacral hiatus in lateral decubitus position after general anesthesia induction. Standard intraoperative monitoring and postoperative care are applied.
  Interventions: Procedure: Caudal epidural block
- Dorsal penile nerve block (Experimental): Participants receive a bilateral dorsal penile nerve block with 0.25% bupivacaine (1 mL/kg divided equally) via the subpubic approach after general anesthesia induction. Standard intraoperative monitoring and postoperative care are applied.
  Interventions: Procedure: Dorsal Penile nerve Block

INTERVENTIONS:
Procedure: Caudal epidural block — A caudal epidural block was performed after induction of general anesthesia with the patient in the lateral decubitus position. A 22-G needle was inserted through the sacral hiatus into the caudal epidural space after loss of resistance of the sacrococcygeal membrane. Bupivacaine 0.25% at a dose of 0.5 mL/kg was injected following negative aspiration.
  Arms: Caudal epidural block
Procedure: Dorsal Penile nerve Block — A dorsal penile nerve block was performed after induction of general anesthesia using the subpubic approach with the patient in the supine position. A 22-G needle was inserted bilaterally at the 10 and 2 o'clock positions near the base of the penis after gentle caudal traction. After negative aspiration, bupivacaine 0.25% at a dose of 1 mL/kg, divided equally on both sides, was injected to block the dorsal penile nerves.
  Arms: Dorsal penile nerve block

SUMMARY:
This prospective, randomized clinical trial conducted at Ain Shams University Hospitals evaluated the analgesic efficacy of dorsal penile nerve block versus caudal epidural block in 30 male children undergoing primary hypospadias repair. Patients were randomly assigned to the penile block group (n=15) or the caudal block group (n=15). Both groups received standardized general anesthesia. The dorsal penile nerve block was performed with 0.25% bupivacaine (1 mL/kg) via a subpubic approach, while the caudal block used 0.25% bupivacaine (0.5 mL/kg) through the sacral hiatus. Block failure was managed with intravenous fentanyl. Baseline demographics and operative duration were comparable between groups. Postoperative pain assessed using the FLACC scale showed superior early analgesia in the caudal group at 0 and 3 hours, with comparable scores at 6-12 hours. The caudal block group required rescue analgesia later and consumed lower total doses of paracetamol and pethidine within 24 hours. However, caudal block delayed ambulation compared to the penile block group. No major complications were reported. The study concludes that both blocks are safe and effective; caudal epidural provides superior early postoperative analgesia, while dorsal penile block may be preferred when early ambulation is desired.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Hypospadias repair remains one of the most common pediatric urological procedures, with thousands of cases performed annually worldwide. Despite continuous refinement of surgical techniques, perioperative pain management in this population poses consistent clinical challenges. Children undergoing hypospadias repair typically experience significant postoperative discomfort due to tissue manipulation, dissection of delicate structures, and exposure of the highly innervated penile shaft. Poorly controlled postoperative pain may lead to increased stress responses, delayed discharge, impaired healing, and difficulties with early postoperative voiding. Because pain expression in young children is complex and often non-verbal, anesthesiologists rely on validated objective scoring systems-such as the FLACC scale-to assess discomfort and guide analgesic therapy.

Regional anesthesia is widely employed as an adjunct to general anesthesia to enhance perioperative analgesia while reducing the need for systemic opioids. Among the most widely used techniques are the caudal epidural block and the dorsal penile nerve block. Each technique has distinct advantages, limitations, and implications for recovery, ambulation, and analgesic duration. Caudal block is traditionally considered the gold standard for infra-umbilical surgeries in pediatrics due to its ease of application, high success rate, and ability to provide profound postoperative analgesia. However, concerns persist regarding delayed motor recovery, urinary retention, and potential adverse hemodynamic effects.

In contrast, the dorsal penile nerve block provides targeted sensory blockade limited to the penile region, minimizing motor involvement and typically allowing earlier mobilization. It is frequently favored in ambulatory settings or when rapid recovery is required. However, its duration of action may be shorter, and there is ongoing debate about whether it can provide analgesic efficacy equivalent to caudal anesthesia following more extensive penile reconstruction, such as hypospadias repair. Given the variation in practice patterns and the lack of high-quality comparative studies in the local setting, this trial was designed to provide a head-to-head comparison of the two regional techniques under standardized anesthetic conditions. The objective was to characterize their intraoperative stability, postoperative pain control, recovery profile, need for rescue analgesia, and safety, enabling clinicians to make informed decisions tailored to patient characteristics, surgical technique, and postoperative care priorities.

STUDY DESIGN OVERVIEW This trial was designed as a prospective, randomized, and comparative clinical study conducted at the Pediatric Surgery Unit of Ain Shams University Hospitals. The study was carried out over a six-month period, following institutional ethical approval, and adhered strictly to the principles of good clinical practice and the Declaration of Helsinki. All participants were recruited consecutively from eligible children scheduled for primary hypospadias repair. A computer-generated randomization sequence was utilized to allocate patients into two equal groups receiving one of two regional anesthesia techniques. All procedures were performed by anesthesiologists with extensive experience in pediatric regional anesthesia, ensuring consistency and proficiency across techniques. A standardized perioperative protocol was applied to all cases to avoid confounding variables. General anesthesia was induced and maintained using identical agents, ventilation strategies, and monitoring parameters. The regional blocks were administered after induction but before surgical incision. Hemodynamic stability, adequacy of analgesia, and possible complications were monitored meticulously throughout the intraoperative and postoperative periods. Data collection continued for the first 24 hours after surgery, with measurements obtained at fixed postoperative intervals. Pain scores, hemodynamic variables, time to ambulation, and need for rescue analgesia were recorded using objective and validated tools. All study staff responsible for postoperative evaluation were blinded to group allocation to minimize assessment bias.

ANESTHETIC MANAGEMENT PROTOCOL A unified anesthetic protocol was implemented for all participants to ensure consistency. Upon arrival in the operating room, each child underwent inhalational induction using 8% sevoflurane in 100% oxygen. Intravenous access was then secured with an appropriately sized cannula (22-24G). Routine monitoring included electrocardiography, non-invasive blood pressure, oxygen saturation, and end-tidal CO₂. Once anesthetized, participants were intubated without the use of neuromuscular blocking agents to prevent interference with motor-based postoperative assessments.

After induction and stabilization, regional anesthesia was performed according to the group assignment. All techniques were executed under sterile conditions using using isoflurane (1-2%) in a mixture of oxygen and air. Ventilation parameters were adjusted to maintain normocapnia. Throughout surgery, continuous monitoring allowed detection of inadequate analgesia. A >20% rise from baseline in mean arterial pressure or heart rate was considered indicative of insufficient block. In such cases, fentanyl 1 µg/kg was administered, and the participant was subsequently excluded from per-protocol analysis to ensure the study accurately reflected the analgesic performance of each regional technique. At the end of surgery, inhalational agents were discontinued, and extubation was performed once all criteria were met, including adequate spontaneous breathing, protective reflexes, and hemodynamic stability. Patients were then transferred to the post-anesthesia care unit (PACU) for initial recovery and postoperative monitoring. DPB is designed to target the primary sensory nerves of the penis at the most proximal location accessible extracorporeally, maximizing analgesic coverage of the penile shaft and glans. It minimizes motor involvement, preserves lower-limb function, and is well suited for early mobilization. Caudal block provides sensory and motor blockade to the lumbosacral dermatomes, ensuring extensive analgesia for penile and perineal surgeries. Its principal advantage is its prolonged analgesic duration, although transient motor impairment may delay ambulation.

PERIOPERATIVE MONITORING AND SAFETY OVERSIGHT

Intraoperative monitoring continued throughout the procedure, with recordings of heart rate, mean arterial pressure, oxygen saturation, and end-tidal CO₂ at predetermined intervals. Any adverse events, such as hypotension, bradycardia, local anesthetic systemic toxicity, arrhythmias, or signs of block-related complications, were documented. Postoperative monitoring focused on detecting pain, hemodynamic alterations, sedation levels, nausea, vomiting, urinary retention, motor impairment, and block-related complications. All assessments were performed in the PACU and continued in the ward at 3, 6, 9, and 12-hour intervals, with additional observations made as clinically necessary. Pain assessment utilized the FLACC scale because of its reliability and effectiveness in non-verbal and preverbal pediatric populations. All nurses and assessors were trained in FLACC scoring to avoid inter-observer variability.

DATA COLLECTION AND MANAGEMENT All collected data, including demographic variables, perioperative measurements, and postoperative findings, were entered into standardized data sheets and subsequently transferred to a secure electronic database. Data accuracy was verified by dual-entry validation. Confidentiality of participant information was strictly maintained, with de-identified codes used for all analyses.

STATISTICAL HANDLING AND ANALYTIC FRAMEWORK Quantitative variables were initially assessed for normality using the Shapiro-Wilk test. Parametric data were analyzed using the independent-samples t-test to compare means between the two groups. Non-parametric variables, including FLACC scores, were analyzed using the Mann-Whitney U test. Categorical variables, such as ASA status, were analyzed using the chi-square test. A 95% confidence interval and significance threshold of p < 0.05 were applied.

STUDY FLOW AND CLINICAL OBSERVATIONS The flow of participants from recruitment through follow-up was documented in accordance with CONSORT guidelines. No block-related complications, such as hematoma, infection, or systemic toxicity, were observed. Both regional techniques demonstrated favorable safety profiles. Clear differences emerged between the two groups in postoperative hemodynamics, pain trajectories, timing of rescue analgesia, and recovery parameters. These findings provided robust comparative insights into the performance of each regional anesthesia modality under consistent surgical and anesthetic conditions.

INTERPRETATION AND CLINICAL SIGNIFICANCE The trial revealed distinct advantages and limitations of each regional technique. Caudal block offered superior early postoperative analgesia and significantly prolonged the time to first analgesic requirement. It also resulted in reduced total consumption of rescue analgesics within 24 hours. These outcomes highlight its value in situations where extended postoperative pain control is a clinical priority. However, the caudal block was associated with delayed ambulation, likely resulting from transient motor involvement in the lower limbs. This consideration is crucial in fast-track surgical settings or when early mobilization is required. The dorsal penile nerve block provided effective analgesia with shorter recovery time and earlier ambulation, making it an appropriate choice for ambulatory care or settings aiming for rapid discharge.

The findings underscore the importance of individualized analgesic planning based on the surgical context, patient characteristics, and recovery goals. Both blocks are safe and effective when performed by skilled practitioners.

CONCLUSION This detailed clinical investigation provides comprehensive comparative data on two widely used regional anesthesia techniques for hypospadias repair. By standardizing anesthetic management, surgical technique, and postoperative assessment, the study establishes strong evidence to guide pediatric pain management and optimize perioperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male children aged 1 to 8 years.
* ASA physical status I or II.
* Scheduled for elective distal or mid-penile hypospadias repair.
* Under general anesthesia.
* Written informed consent obtained from parents or legal guardians.

Exclusion Criteria:

* Age < 1 year or > 8 years.
* ASA physical status III or higher.
* Complicated hypospadias.
* Coagulopathy or ongoing anticoagulant therapy.
* Known allergy or contraindication to local anesthetics.
* Significant neurological or neuromuscular disorders affecting pain perception.
* Vertebral anomalies.
* Local infection at the site of injection.
* Refusal or inability of parents/guardians to provide informed consent.

Ages: 1 Year to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesia. | Within the first 24 hours postoperatively
  Time elapsed from the end of surgery until the first administration of rescue analgesia.
Total 24-hrs postoperative analgesic consumption. | Within the 24 hours postoperatively
  Total amount of postoperative analgesics (paracetamol and pethidine) administered during the first 24 hours after surgery, expressed as mg/kg.

SECONDARY OUTCOMES:
Postoperative Pain Score using Face, Legs, Activity, Cry, Consolability ( FLACC score) | At PACU, and 3, 6, 9, and 12 hours postoperatively.
  Pain intensity will be assessed using the Face, Legs, Activity, Cry, Consolability (FLACC) scale, which ranges from 0 (no pain) to 10 (worst possible pain), with higher scores indicating more severe pain.
Time to Ambulation | Within the first 24 hours postoperatively
  Time from the end of surgery until the patient was able to ambulate.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam K Habib, MD, Principal Investigator — Ain Shams University
Locations (1):
- intensive care unit Department, Ain Shams University Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) including age, weight, ASA status, FLACC scores, and analgesic consumption will be shared with qualified researchers upon request after publication. Requests will be reviewed by the Principal Investigator, and approved data will be shared via a secure repository. No personal identifiers will be included.
Supporting Information: SAP, CSR
Time Frame: Start Date: Upon publication of the study results. End Date: 5 years after publication.
Access Criteria: Qualified researchers who provide a methodologically sound proposal and have obtained approval from the study investigators will be able to access the de-identified individual participant data and relevant supporting documents. Requests should be submitted via email to the corresponding author, and data will be shared under a data use agreement ensuring confidentiality and proper use.